CLINICAL TRIAL: NCT04652817
Title: An Open-Label Uncontrolled Single Centre Study for the Evaluation of the Performance Characteristics (Efficacy and Safety) of the Dermal Filler MMI-22-04-2019 (Hyaluronic Acid 2,5%) for Female Intimate Area Augmentation of Labia Majora.
Brief Title: Evaluation of the Efficacy and Safety of the Dermal Filler for Augmentation of Labia Majora.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD/MMI-22-04-2019
Record Dates: First submitted 2020-02-20; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Labia Majora Atrophy and Hypotrophy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MMI-22-04-2019 (Experimental): Sodium hyaluronate at a concentration of 2.5% (25 mg/ml) with 1,4-Butanediol diglycidyl ether (BDDE) acting as a cross-linking agent administered once or twice depending on the individual necessity.
  Interventions: Device: MMI-22-04-2019

INTERVENTIONS:
Device: MMI-22-04-2019 — A cross-linked form of the Hyaluronic Acid is used in intradermal injection to augment the labia majora area.

SUMMARY:
The study is an open-label uncontrolled single-center study for the evaluation of the Performance characteristics (efficacy and safety) of the dermal filler "MMI-22-04-2019" on the female genital area for the aesthetic, medicinal, functional and reconstructive indications.

DETAILED DESCRIPTION:
MMI-22-04-2019 is a dermal filler recommended for application in the intimate area. It is a sterile, injectable, colorless transparent gel, non-pyrogenic, reabsorbable medical device. Its main functional ingredient is cross-linked hyaluronic acid of non-animal origin, produced through bacterial fermentation.

The MMI-22-04-2019 is contained in pre-filled, graduated, disposable sterile syringe with Luer Lock adapter with 1 ml of net content. The sterilization of the product is achieved by moist heat.

The MMI-22-04-2019 has been classified as a Class III medical device under Annex IX of Directive MDD 93/42 EEC since it is a long-term, invasive and absorbable medical device.

ELIGIBILITY:
Inclusion Criteria:

* Female subject aged ≥18;
* Subject presenting vulvar ptosis, deflation or aesthetic discomfort in the intimate area;
* Subject who presents no type of pathology of the area to be treated;
* Subjects who are willing to abstain from any cosmetic or surgical procedures in the treatment area during the clinical investigation;
* Clinically and anamnestically healthy individual;
* Absence of a history of significant hypersensitivity to food and drugs or known sensitivity to hyaluronic acid;
* Arterial blood pressure (BP) (after 5 min. at rest in the supine position) systolic 90 - 140 mmHg and diastolic 50 - 90 mmHg;
* Heart rate (HR) (after 5 min. at rest in the supine position) over 50 beats/min and less than 90 beats/min;
* Respiratory rate between 12 - 24 breaths/min;
* Axillar body temperature of up to 370С;
* Clinical-laboratory examinations within the reference ranges or with no clinically significant abnormalities;
* Negative AIDS/HIV test;
* Negative pregnancy test for the women with reproductive potential;
* Reliable and acceptable method of contraception for the women of child-bearing potential
* Signed written Informed Consent Form.

Exclusion Criteria:

* Subject with known sensitivity to hyaluronic acid or significant hypersensitivity to food and drugs;
* Subject with history of vulvar cancer and/or previous regional radiotherapy;
* Subjects with frequent or present active herpes simplex or herpes zoster local infection or active herpes simplex or herpes zoster infection in other sites;
* Subjects with history of frequent or active local dermatitis (of the injection site), vulvar scaly papilloma, mycosis; bacterial infection;
* Subjects suffering from autoimmune diseases or who are undergoing treatment with immunosuppressors or immunotherapy;
* Subjects uncontrolled systemic diseases;
* Pregnancy, postpartum period (6 months) or post-lactation period (6 months);
* Absence of a reliable and effective method of contraception;
* Subjects who are currently receiving another investigational treatment or who had participated in another clinical investigation within 30 days prior to study enrollment;
* Subjects who suffer from another medical condition or who are receiving medication that in the Principal Investigator's judgment would prohibit inclusion in the study;
* Subjects with limited mental activity and consistent comprehension ability; sportsmen and individuals on strenuous physical loading; prisoners;
* Refusal to sign the Informed Consent Form.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender-based pathology.
Enrollment: 35 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Visual Analogous Scale (VAS) absolute change | From Day 0 (Session 1) to Day 60 (Session 3) - up to 8 weeks.
  The absolute change in VAS, judged by the Principal Investigator. VAS ranged between 0 (least satisfied) and 10 (most satisfied) is used. The higher the score, the better the cosmetic appearance.
Treatment-Emergent Adverse Events [Safety and Tolerability] | From screening through study completion, an average of 90 days - daily.
  Frequency and severity of adverse events (AEs) and adverse device effects.

SECONDARY OUTCOMES:
Visual Analogous Scale (VAS) | From Day 0 (Session 1) to Day 0 (immediately after application), 30 (up to 4 weeks) and 90 (up to 12 weeks) (Session 1, 2 and 4).
  The absolute change in VAS, judged by the Principal Investigator. VAS ranged between 0 (least satisfied) and 10 (most satisfied) is used. The higher the score, the better the cosmetic appearance.
Global Aesthetic Improvement Scale (GAIS) | From Day 0 (immediately after application) to Days 30, 60 and 90 (up to 4 weeks, 8 weeks and 12 weeks respectively).
  The change in GAIS as evaluated by the PI based on the photographs of the treated area. A 5-point scale rating improvement in appearance compared to pre-treatment - 1 being exceptional improvement and 5 being worsened.
Subject satisfaction | Days 0 (immediately after application), 30, 60 and 90 (up to 4 weeks, 8 weeks and 12 weeks respectively).
  Subject satisfaction based on Questionnaire, including visual analogue scale, ranged between 0 (least satisfied) and 10 (most satisfied) is used and questions about discomfort and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Ramus, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No